CLINICAL TRIAL: NCT06724211
Title: Preventing Delayed Graft Function in Kidney Transplant Patients: A Single-centre, Randomised, Feasibility Trial
Brief Title: Preventing Delayed Graft Function in Kidney Transplant Patients
Acronym: PDF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 24-5286
Record Dates: First submitted 2024-11-26; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplant; Kidney Failure; Kidney Injury
Keywords: Kidney Transplant; Surgical Bundle
MeSH Terms: conditions — Renal Insufficiency | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either the experimental group, which will consist of a treatment bundle of care, or to the control group, which will consist of routine clinical care for kidney transplant patients. The treatment bundle of care will consist of: the use of plasmalyte for fluid management, maintaining mean arterial pressure > 75 mmHg, identify and treat blood glucose > 9 mmol/L, and a restrictive criteria for red blood cell transfusions (i.e. hemoglobin (Hb) < 70 g/L).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Routine clinical care for kidney transplant patients
  Interventions: Other: Control Group
- Surgical bundle (Experimental): The surgical bundle will consist of: the use of plasmalyte for fluid management, maintaining mean arterial pressure > 75 mmHg, identify and treat blood glucose > 9 mmol/L, and a restrictive criteria for red blood cell transfusions (i.e. hemoglobin (Hb) < 70 g/L).
  Interventions: Other: Treatment bundle of care

INTERVENTIONS:
Other: Treatment bundle of care — The treatment bundle of care will consist of: the use of plasmalyte for fluid management, maintaining mean arterial pressure > 75 mmHg, identify and treat blood glucose > 9 mmol/L, and a restrictive criteria for red blood cell transfusions (i.e. hemoglobin (Hb) < 70 g/L).
  Arms: Surgical bundle
Other: Control Group — Routine clinical care for kidney transplant patients
  Arms: Control Group

SUMMARY:
The health and quality of life benefits of kidney transplantation are reduced by delayed graft function (DGF). There are a number of modifiable risk factors associated with DGF, such as intraoperative hypotension, the type of intravenous fluid used, glycemic control, and the restriction of blood transfusions. However, these factors have been assessed individually, and their collective effect on reducing the risk of DGF requires further investigation. We first propose a pilot RCT to establish the feasibility of a definitive RCT examining the impact of a treatment bundle of care on DGF.

This will be a single centre, double-blinded pilot RCT including 50 adults undergoing kidney transplantation. Patients will be randomized to either the experimental group, which will consist of a treatment bundle of care, or to the control group, which will consist of routine clinical care for kidney transplant patients. The treatment bundle of care will consist of: the use of plasmalyte for fluid management, maintaining mean arterial pressure > 75 mmHg, identify and treat blood glucose > 9 mmol/L, and a restrictive criteria for red blood cell transfusions (i.e. hemoglobin (Hb) < 70 g/L).

The primary outcome of this pilot study is the recruitment rate. Recruitment rate will be defined as the number of patients who are approached to participate in the study and who are randomized to either the experimental or control group, as a percentage of the total number of eligible kidney transplant patients. The secondary outcomes are: 1) protocol adherence rate and 2) follow-up rate. Protocol success will be defined as a ≥90% compliance with at least 3 of the 4 treatment bundle components. Patient follow-up will end at 90-days after transplant and the target is to follow ≥90% of the patients until this time. DGF and acute rejection will not be assessed in the feasibility trial, and instead this data will be analyzed in the full trial.

DETAILED DESCRIPTION:
Background: A number of perioperative factors can impact graft function after kidney transplant, such as hypotension, type of intravenous fluid used, red blood cell transfusions and glycemic control. For example, we recently found that intraoperative hypotension was associated with DGF-CRR following kidney transplant, with a threshold mean arterial blood pressure of 65 mmHg (manuscript submitted). Furthermore, the odds of DGF-CRR increased when the MAP was < 75 mmHg. A method to manage blood pressure during kidney transplant is administering intravenous fluids, either with crystalloids or blood. A recent multicenter, randomized controlled trial showed that plasmalyte, a balanced crystalloid fluid, reduces the incidence of DGF-D after DD- kidney transplant by 25% (i.e. 40% to 30%) compared to normal saline. In the kidney transplant population, blood transfusion was reported to be associated with reduced graft function, early graft loss, and reduced patient survival. As the vast majority of patients receiving blood transfusion receive only 1-2 units, many transfusion events likely could be avoided with better adherence to appropriate triggers, potentially leading to improved outcomes following kidney transplant. Finally, irrespective of a pre-transplant diabetes diagnosis, hyperglycemia (blood sugar > 9.0 mmol/L) in the post-anesthesia care unit is associated with an increased odds of DGF-D following kidney transplant. Therefore, glucose control (i.e. blood sugar < 9 mmol/L) may improve immediate graft function in this patient population.

Rationale: Preserving graft function following kidney transplant is critical to ensuring favourable outcomes. We propose to study the application of a modified version of the KDIGO guidelines for kidney transplant patients. This perioperative bundle of care includes maintenance of MAP >75 mmHg after kidney reperfusion, use of plasmalyte for fluid administration, reducing red blood cell transfusion and identifying and treating a blood sugar > 9 mmol/L. Although this care bundle shows promise for reducing the risk of DGF following transplant, this should first be investigated in a pilot, feasibility trial to ensure successful patient recruitment and adherence to the study protocol, prior to undergoing a full RCT.

Hypothesis: We hypothesize that the proposed perioperative bundle of care will be feasible to implement and improve postoperative outcomes for kidney transplant recipients.

Primary Objectives: The primary objective is to determine the feasibility of recruiting and randomizing kidney transplant recipients to an RCT evaluating the administration of a perioperative bundle of care. Recruitment rate will be defined as the number of patients who are approached to participate in the study and who are randomized to either the treatment or routine clinical care group, as a percentage of the total number of eligible transplant patients. In order to complete a full multicenter trial in a reasonable time period (2-3 years), the number needed to recruit per week is at least 1 patient, but we will aim to recruit 2 patients per week.

The secondary objective is to determine protocol adherence and follow-up rates. The aim is for ≥90% compliance with at least 3 of the 4 components of the perioperative bundle of care i.e. use of Plasmalyte for fluid management, maintenance of MAP > 75 mmHg from time of cross-clamp removal to 4-hours post KT, the initiation of an insulin infusion to maintain a serum blood sugar < 9 mmol/L and avoidance of RBC transfusion unless the Hb < 70 g/L or symptoms of oxygen insufficiency and Hb < 80 g/L. For this trial, patient follow-up will end at 90-days after transplant and the target is to follow ≥90% of the patients until this time. DGF and acute rejection will not be assessed in the feasibility trial, and instead this data will be analyzed in the full trial. Patient follow-up of clinical outcomes will occur at 1-year following KT in the full trial.

Study Significance: This pilot study seeks to assess whether we can recruit kidney transplant patients for an RCT and assess compliance to a surgical care bundle aiming to reduce the incidence of delayed graft function. Preserving graft function after transplant is critical to ensuring favourable outcomes. The primary objectives of this study will assess protocol adherence and outcome collection rates. The results of this pilot trial will serve as the rationale to conduct a large, randomized controlled trial with the use of the surgical care bundle to enhance the recovery of kidney transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Patients undergoing kidney transplantation
* Living and deceased donor recipients

Exclusion Criteria:

* Multi-organ transplant
* Pre-emptive KT
* Arterial line not planned for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline, pre-intervention/procedure/surgery
  Recruitment rate will be defined as the number of patients who are approached to participate in the study and who are randomized to either the treatment or routine clinical care group, as a percentage of the total number of eligible transplant patients.
  In order to complete a full multicenter trial in a reasonable time period (2-3 years), the number needed to recruit per week is at least 1 patient, but we will aim to recruit 2 patients per week.

SECONDARY OUTCOMES:
Protocol adherence | During the intervention/procedure/surgery AND immediately after the intervention/procedure/surgery
  The aim is for ≥90% compliance with at least 3 of the 4 components of the perioperative bundle of care i.e. use of Plasmalyte for fluid management, maintenance of MAP > 75 mmHg from time of cross-clamp removal to 4-hours post KT, the initiation of an insulin infusion to maintain a serum blood sugar < 9 mmol/L and avoidance of RBC transfusion unless the Hb < 70 g/L or symptoms of oxygen insufficiency and Hb < 80 g/L.
Follow-up rate | 90-days after final patient recruited
  Patient follow-up will end at 90-days after transplant and the target is to follow ≥90% of the patients until this time. DGF and acute rejection will not be assessed in the feasibility trial, and instead this data will be analyzed in the full trial. Patient follow-up of clinical outcomes will occur at 1-year following KT in the full trial.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Dr. McCluskey, MD, PhD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Sharing such detailed data can risk exposing sensitive personal information, even if anonymized. Additionally, there are often ethical and legal considerations that restrict the sharing of IPD to protect participants' rights and comply with regulations.

REFERENCES:
- [Result] Sicova M, McGinn R, Emerson S, Perez P, Gonzalez R, Li Y, Famure O, Randall I, Mina DS, Santema M, Wijeysundera DN, Van Klei W, Kim SJ, McCluskey SA. Association of Intraoperative Hypotension With Delayed Graft Function Following Kidney Transplant: A Single Centre Retrospective Cohort Study. Clin Transplant. 2024 Oct;38(10):e70000. doi: 10.1111/ctr.70000. PMID 39460628
- [Result] Pascoe EM, Chadban SJ, Fahim MA, Hawley CM, Johnson DW, Collins MG; BEST-fluids Investigators and the Australasian Kidney Trials Network. Statistical analysis plan for Better Evidence for Selecting Transplant Fluids (BEST-Fluids): a randomised controlled trial of the effect of intravenous fluid therapy with balanced crystalloid versus saline on the incidence of delayed graft function in deceased donor kidney transplantation. Trials. 2022 Jan 18;23(1):52. doi: 10.1186/s13063-021-05989-w. PMID 35042554

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT06724211/Prot_SAP_000.pdf